CLINICAL TRIAL: NCT04973033
Title: Tofacitinib for the Treatment of Anti-Neutrophil Cytoplasm Antibody-associated Vasculitis: a Pilot Study
Brief Title: Effect of Tofacitinib in Treating ANCA-associated Vasculitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TofAV
Record Dates: First submitted 2021-07-05; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: ANCA Associated Vasculitis; Drug Use; JAK-STAT Pathway Deregulation
Keywords: ANCA associated vasculitis; tofacitinib; safety; efficacy
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — tofacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tofactitinib (Experimental): Tofacitinib 5mg twice a day
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — patients enrolled were prescribed tofacitinib 5mg twice a day orally.
  Other Names: Tofacitinib 5mg.bid.po.

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of tofacitinib 5 mg twice daily in AAV patients.

DETAILED DESCRIPTION:
Anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV) represents a group of small vessel vasculitides characterized by granulomatous and neutrophilic tissue inflammation, often associated with the production of antibodies that target neutrophil antigens. The predominantly used treatment for induction of remission in AAV consisted of cyclophosphamide (CYC) plus corticosteroids (GCs) which leads to remission in about 90% of patients. However, relapses are frequent and remain a challenge. The optimal drug for maintenance treatment is not determined. Tofacitinib is a Jak inhibitor which has been proved to be effective in multiple inflammatory diseases such as rheumatoid arthritis. Considering that T cells and associated cytokine production play an important role in the pathogenesis of AAV via activation of the JAK/ STAT pathway, we hypothesized that tofacitinib-mediated inhibition of JAK signaling may represent an effective therapy for active AAV. In this prospective, open label, single arm study, tofacitinib 5mg twice a day will be added to the background treatment of GCs and immunosuppressants in AAV, the safety and efficacy of tofacitinib will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active AAV met the criteria of 1990 ACR and 2012 Chapel Hill criteria
* Age 18 to 75 years
* Written informed consent obtained before taking part in the study

Exclusion Criteria:

* Severe AAV defined as potentially organ- or life-threatening disease (i.e. alveolar haemorrhage, heart failure caused by myocarditis or pericarditis, progressive neurological symptoms, deaf, blindness, et al.)
* Serum creatinine>120umol/L or proteinuria>1.0g/d
* Receipt of a JAKi therapy previously
* Co-existence of another systemic autoimmune disease
* Secondary vasculitis (following neoplastic disease, an infection or antithyroid drugs)
* Malignancy or history of malignancy
* Infection by HIV, HCV, HBV or tuberculosis-
* Severe uncontrolled cardiovascular, pulmonary, liver, gastrointestinal, endocrine, hematological, neurological, or psychiatric diseases that are not related to systemic vasculitis
* Allergic to JAKi
* Blood dyscrasias including confirmed: Hemoglobin <9 g/dL or Hematocrit <30%; White blood cell count <3.0 x 109/L; Absolute neutrophil count <1.5 x 109/L; Platelet count <100 x 109/L; Alanine transaminase or aspartate aminotransferase or total bilirubin>1.5 upper normal limit; Estimated glomerular filtration rate<60ml/min/1.73m2
* Incapacity or refusal to understand or sign the informed consent form.
* Pregnancy, breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
The response rate (CR, PR and TR) | From the enrollment to the end of follow-up [0 to 13 months.]
  The percent of patients who achieved disease response. The disease response includes:(1) complete remission (CR), defined as the absence of disease activity (BVAS = 0); (2) partial remission (PR) defined as at least 50% reduction of BVAS and no new manifestations; (3) treatment resistance (TR) was defined as less than a 50% reduction or increased disease activity after 4 ~ 6 weeks of treatment.

SECONDARY OUTCOMES:
The rate of adverse event | From the enrollment to the end of follow-up [0 to 13 months].
  The percent of different kinds of adverse events occurred during follow-up. The adverse event was evaluated according to the CTC-AE 4.0 standard.
Changes in erythrocyte sedimentation rate (ESR) | From the enrollment to the end of follow-up [0 to 13 months].
  The change of ESR in different follow-up point compared with the baseline.
Changes in CRP | From the enrollment to the end of follow-up [0 to 13 months].
  The change of CRP in different follow-up point compared with the baseline.
Changes in glucocorticoids steroids (GCs) dosage | From the enrollment to the end of follow-up [0 to 13 months].
  The change of the prednisone or its equivalent drug in different follow-up point compared with the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Lindi Jiang, PhD, Study Chair — Fudan University
Locations (1):
- Department of Rheumatology in Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality, China